CLINICAL TRIAL: NCT03007875
Title: High-activity Natural Killer Immunotherapy for Small Metastases of Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HANK-nsclc
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2018-12

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: Metastatic lung cancer; High-activity natural killer
MeSH Terms: conditions — Lung Neoplasms

ARMS (2):
- High-activity natural killer (Experimental): In this group, the patients will receive multiple times of high-activity natural killer (HANK) immunotherapies. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Biological: high-activity natural killer
- ControL (No Intervention): In this group, the patients will receive no special treatment and as a control group. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).

INTERVENTIONS:
Biological: high-activity natural killer — Each treatment: 8~10 billion cells in all, transfuion in 3 times, i.v.
  Other Names: HANK cell
  Arms: High-activity natural killer

SUMMARY:
The aim of this study is the safety and efficacy of high-activity natural killer immunotherapy to small metastases of non-small cell lung cancer.

DETAILED DESCRIPTION:
By enrolling patients with small metastases of non-small cell lung cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of high-activity natural killer cells.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 2 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Relief degree of tumors | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Overall survival（OS） | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fuda cancer institute of Fuda cancer hospital, Guangzhou, Guangdong, China